CLINICAL TRIAL: NCT02758405
Title: Programmed Intermittent Epidural Bolus for Labor Analgesia During First Stage of Labor: A Sequential Allocation Trial to Determine the Optimum Interval Time Between Boluses of a Fixed Volume of 5 of Bupivacaine 0.125% Plus Fentanyl 2 mcg/ml.
Brief Title: Programmed Intermittent Epidural Bolus for Labor Analgesia During First Stage of Labor 2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samuel Lunenfeld Research Institute, Mount Sinai Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 16-03
Record Dates: First submitted 2016-04-29; First posted 2016-05-02 (Estimated); Last update posted 2017-05-24 (Actual); Status verified 2017-05

CONDITIONS: Labor Pain
Keywords: Epidural; Labor analgesia; Programmed intermittent epidural bolus
MeSH Terms: conditions — Labor Pain | interventions — Bupivacaine; Fentanyl; Infusion Pumps

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- 60 minutes (Experimental): The infusion pump will deliver programmed intermittent epidural boluses at a 60-minute interval. The bolus will consist of 5mL of 0.125% Bupivacaine plus fentanyl 2mcg/ml. A PCEA bolus of 5mL of 0.125% Bupivacaine plus fentanyl 2mcg/ml will also be available.
  Interventions: Drug: Bupivacaine; Drug: Fentanyl; Device: Infusion pump
- 50 minutes (Experimental): The infusion pump will deliver programmed intermittent epidural boluses at a 50-minute interval. The bolus will consist of 5mL of 0.125% Bupivacaine plus fentanyl 2mcg/ml. A PCEA bolus of 5mL of 0.125% Bupivacaine plus fentanyl 2mcg/ml will also be available.
  Interventions: Drug: Bupivacaine; Drug: Fentanyl; Device: Infusion pump
- 40 minutes (Experimental): The infusion pump will deliver programmed intermittent epidural boluses at a 40-minute interval. The bolus will consist of 5mL of 0.125% Bupivacaine plus fentanyl 2mcg/ml. A PCEA bolus of 5mL of 0.125% Bupivacaine plus fentanyl 2mcg/ml will also be available.
  Interventions: Drug: Bupivacaine; Drug: Fentanyl; Device: Infusion pump
- 30 minutes (Experimental): The infusion pump will deliver programmed intermittent epidural boluses at a 30-minute interval. The bolus will consist of 5mL of 0.125% Bupivacaine plus fentanyl 2mcg/ml. A PCEA bolus of 5mL of 0.125% Bupivacaine plus fentanyl 2mcg/ml will also be available.
  Interventions: Drug: Bupivacaine; Drug: Fentanyl; Device: Infusion pump

INTERVENTIONS:
Drug: Bupivacaine — 0.125% Bupivacaine plus fentanyl 2mcg/ml
  Other Names: Marcaine
Drug: Fentanyl — 0.125% Bupivacaine plus fentanyl 2mcg/ml
Device: Infusion pump — Infusion pump set to deliver programmed intermittent epidural boluses (PIEB) plus patient-controlled epidural analgesia (PCEA).
  Other Names: CADD-Solis Ambulatory Infusion Pump

SUMMARY:
Brief Summary:

Until recently, at Mount Sinai Hospital, epidural analgesia for labor pain was delivered with a pump that could only provide continuous infusion of the freezing medication in combination of pushes of medication activated by the patient, a technique called patient controlled epidural analgesia (PCEA). In the last decade or so, the literature has suggested that this continuous infusion of medication is not as effective as previously thought, and suggested that instead of continuous infusion, intermittent programmed pushes should be used. The investigators now have devices that are able to do that. Programmed intermittent epidural bolus (PIEB) is a new technological advance based on the concept that boluses of freezing medication in the epidural space are superior to continuous epidural infusion (CEI). The investigators are currently using pumps set up with PIEB, in addition to what the patient can deliver herself (PCEA). Studies have shown that delivering analgesia in this manner prolong the duration of analgesia, reduce motor block, lower the incidence of breakthrough pain, improve maternal satisfaction and decrease local anesthetic consumption. The investigators have recently concluded a study at MSH using PIEB where they observed excellent results. However, some patients exhibited higher than necessary sensory blocks. The investigators believe that the technique can be optimized by using the same dose of the freezing medication, but using a smaller volume of local anesthetic at a higher concentration. This optimization may also further reduce the amount of medication used by each patient.

The hypothesis of this study is that there is an optimal interval time between PIEB boluses of 30 to 60 minutes at a fixed volume of 5 ml of bupivacaine 0.125% with fentanyl 2mcg/ml that will provide women the necessary drug requirements, thus avoiding breakthrough pain and need for PCEA or physician intervention.

DETAILED DESCRIPTION:
Studies involving programmed intermittent epidural bolus (PIEB) to date have provided an analgesic regimen that delivered an amount of local anesthetic that was below the patient's requirement per hour, as the studies were done in the context of an association with patient controlled epidural anesthesia (PCEA) as a rescue technique. As a result, PCEA requests were frequent and therefore these studies have not been able to truly understand the pharmacology of the bolus technique in the PIEB regimen, as the PCEA utilized by patients added an extra component to the regimen.

At Mount Sinai Hospital, PIEB devices have been recently introduced. Currently our standard epidural mixture is bupivacaine 0.0625% with fentanyl 2mcg/ml. Based on previous research done by the investigators, the current epidural regimen consists of 10 ml PIEB at 40 minute intervals, with PCEA boluses of 5 ml and a lock out interval of 10 minutes, for a maximum of 20 ml of the epidural mixture per hour.

In this study, the investigators will offer patients 5mL PIEBs of bupivacaine 0.125% with fentanyl 2mcg/ml at 4 different intervals. PCEA bolus of 5mL of the same solution will also be available. The goal is to establish the ideal PIEB regimen that will be effective for our patient population using a higher concentration epidural mixture.

ELIGIBILITY:
Inclusion Criteria:

* ASA 2 or 3
* Full term (≥ 37 weeks gestation)
* Nulliparous
* Singleton pregnancy, vertex presentation
* Active labor: regular painful contractions occurring at 3-at least every 5 minutes and change in cervix
* Verbal Numerical Pain Score (VNPS) at requesting analgesia > 5 (VNPS 0-10)
* Cervical dilatation ≥2 ≤ 5 cm

Exclusion Criteria:

* Refusal to provide written informed consent.
* Any contraindication to epidural anesthesia
* Unintentional dural puncture
* Allergy or hypersensitivity to bupivacaine or fentanyl
* Use of opioids or sedatives within the last 4 hours.

Ages: 16 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2016-05; Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Adequate response of the patient, defined as no request for supplemental analgesia | 6 hours
  Adequate response of the patient, defined as no request for supplemental analgesia (PCEA bolus or clinician administered bolus) until the completion of the first stage of labor or until 6 hours following initiation of the programmed intermittent epidural bolus (PIEB).

SECONDARY OUTCOMES:
Sensory block level | 6 hours
  Sensory block to ice will be assessed bilaterally at the mid axillary lines, and the level of block will be the level at which the patient still does not feel cold sensation as compared to a control site (frontal part of the head)
Motor block level assessed using Bromage score | 6 hours
  Motor block will be assessed with the Bromage score: 0 = able to raise the extended leg; 1 = unable to raise the extended leg but able to flex knees; 2 = unable to flex knees, but able to flex ankle; 3 = unable to flex ankle.
Hypotension | 6 hours
  A decrease in systolic blood pressure greater than 20% from baseline (defined as an average of 3 readings prior to epidural).
Pain score | 6 hours
  Pain score measured hourly using VNRS (0-10)

CONTACTS AND LOCATIONS:
Overall Officials: Jose CA Carvalho, MD, Principal Investigator — MOUNT SINAI HOSPITAL
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No